CLINICAL TRIAL: NCT01120782
Title: Non-dispensing Study to Check Prescription Equivalence of Two Daily Disposable Toric Contact Lens Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-1476AI
Record Dates: First submitted 2010-05-04; First posted 2010-05-11 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-09

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- etafilcon A toric new lens/etafilcon A toric lens (Active Comparator): The lens worn first is a new etafilcon A toric contact lens and the lens worn second is a marketed etafilcon A toric contact lens. Each lens worn for a maximum of 15 minutes bilaterally.
  Interventions: Device: etafilcon A toric contact lens with new wetting agent; Device: etafilcon A toric contact lens
- etafilcon A toric lens/etafilcon A toric new lens (Active Comparator): The lens worn first is a marketed etafilcon A toric contact lens and the lens worn second is a new etafilcon A toric contact lens. Each lens worn for a maximum of 15 minutes bilaterally.
  Interventions: Device: etafilcon A toric contact lens with new wetting agent; Device: etafilcon A toric contact lens

INTERVENTIONS:
Device: etafilcon A toric contact lens with new wetting agent — Investigational toric contact lens made of etafilcon A material with a new wetting agent.
Device: etafilcon A toric contact lens — Marketed toric contact lens made of etafilcon A material.

SUMMARY:
The purpose of this study is to determine whether the prescription determined for a new daily disposable toric contact lens will be a good match to a prescription determined for an existing brand of lens.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be between 18 and 40 years old.
2. The subject must have normal eyes.
3. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
4. The subject must read and sign the STATEMENT OF INFORMED CONSENT and be provided a copy of the form.
5. The subject must have a subjective distance spectacle prescription in the range of -1.75 to -5.00 DS in each eye.
6. The subject must manifest -1.25 to -2.00 D of refractive astigmatism in each eye.
7. The subject's refractive cylinder axis must be 180 +/- 30 in each eye.
8. The subject must be an adapted wearer of soft toric contact lenses in both eyes.
9. The subject's best visual acuity (BVA) must be better than or equal to 20/25 in each eye.
10. Subjects must already possess a wearable pair of spectacles. -

Exclusion Criteria:

1. Ocular or systemic allergies or disease that may interfere with contact lens wear.
2. Systemic disease or autoimmune disease or use of medication, which may interfere with contact lens wear.
3. Clinically significant corneal edema, corneal vascularization, corneal staining or any other abnormality of the cornea, which may contraindicate contact lens wear.
4. Clinically significant tarsal abnormalities that might interfere with contact lens wear.
5. Any ocular infection.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Pregnancy or lactation
8. Any infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
9. Diabetes
10. Strabismus -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-02-01 (Actual); Study Completion 2010-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jacksonville, Florida
  - New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to test article shipment error, one clinical site did not receive control test article in a required cylinder and all screened/enrolled subject were unable to be fitted according to the protocol and were discontinued.
Groups:
- All Subjects: All subjects wore both the test and control lenses: etafilcon A toric contact lens with a new wetting agent and the marketed etafilcon A toric contact lens. Each lens was worn for a maximum of 15 minutes bilaterally.
Period: Overall Study
Arm/Group | All Subjects
Started | 45
Completed | 34
Not Completed | 11
Not completed — Test article shipping error | 11

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (5.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Prescription Equivalence
Description: Number of subjects whose prescription is the same for the two lenses tested.
Time Frame: after 15 minutes of lens wear
Population: All completed subjects.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 34
participants | 34

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires agreement and written authorization from Sponsor.